CLINICAL TRIAL: NCT04169087
Title: Validation and Clinical Implications of the Korean Version of the "Quality of Recovery 15" After General Anesthesia: A Prospective Observational Cohort Study
Brief Title: Korean Version of the "Quality of Recovery 15" After General Anesthesia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: HS-2019-02
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia: Patients undergoing general anesthesia
  Interventions: Other: QoR-15

INTERVENTIONS:
Other: QoR-15 — The QoR-15 is the questionnaire to provide an evaluation of the postoperative quality of recovery. Patients undergoing surgery and general anesthesia are asked by the investigators to complete the QoR-15 questionnaire before and 24h after the surgery.

SUMMARY:
The aim of this study is to test the Korean version of QoR-15 for its validity and clinical acceptability and feasibility.

DETAILED DESCRIPTION:
Quality of recovery (QoR) after anesthesia is an important measure of the early postoperative health status of patients. The QoR-40 is a widely-used questionnaire for postoperative patients and the short-form version of it (QoR-15) was developed in 2013. The validation of QoR-15 has been reported in the version of English, Portuguese, Danish, Chinese and Swedish. However, the study to validate the Korean version of QoR-15 has not been demonstrated.

Patients undergoing surgery and general anesthesia are asked by the investigators to complete the QoR-15 questionnaire and Korean 36-Item Short Form Health Survey (SF-36) a day before surgery. They are then asked to repeat the QoR-15 questionnaire 24 h postoperatively and also rate their overall postoperative pain score using 11-point numeric rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective general surgery, thoracic surgery and gynecological surgery under general anesthesia
* Age between 18 and 80 years
* Willingness and ability to sign an informed consent document
* Ability to understand the contents of questionnaires

Exclusion Criteria:

* Age under 18 or over 80.
* Do not understand our study
* Medical or psychological disease that can affect the treatment response

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery and general anesthesia in Seoul National University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Convergent Validity of the QoR (Quality of Recovery)-15 | 24 hours after the surgery
  The QoR-15 (0-150) is compared with the global QoR visual analog scale (VAS) (0-100), 36-Item Short Form Health Survey (SF-36) and interitem correlations are measured.
Construct Validity of the QoR (Quality of Recovery)-15 | 24 hours after the surgery
  To investigate if there is an correlation between the QoR-15 (0-150) and age (yr), gender (male/female), American Society of Anesthesiologists (ASA) physical status (I-IV), type of surgery (minor/major), postoperative complication (Clavien Dindo grade II or high, %) and 11-point numeric rating scale (NRS) pain score.
Discriminant Validity of the QoR (Quality of Recovery)-15 | 24 hours after the surgery
  To investigate if there is differences in the QoR-15 (0-150) and postoperative complications (Clavien Dindo grade II or high, %) between the high QoR score group and low QoR score group

SECONDARY OUTCOMES:
Reliability of the QoR (Quality of Recovery)-15 | 24 hours after the surgery
  Compare the two QoR-15 results measured at 60 minutes intervals using an intraclass correlation coefficient, and calculate the Cronbach alpha to investigate the internal consistency.
Response success rate of the QoR-15 | A day before and 24 hours after the surgery
  Defined as success if the patient has answered all items.
Correlation of postoperative outcomes with QoR-15 | 24 hours after the surgery
  To investigate if there is an correlation between the QoR-15 (0-150) at POD1 and length of hospital stay (day), postoperative complications (Clavien Dindo grade II or high, %), C-reactive protein (mg/L) at POD1, Granulocyte/lymphocyte ratio at POD1, readmission rate within 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Result] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Derived] Yoon S, Joo H, Oh YM, Lee J, Bahk JH, Lee HJ. Validation and clinical utility of the Korean version of the Quality of Recovery-15 with enhanced recovery after surgery: a prospective observational cohort study. Br J Anaesth. 2020 Oct;125(4):614-621. doi: 10.1016/j.bja.2020.06.040. Epub 2020 Jul 21. PMID 32703550